CLINICAL TRIAL: NCT01468740
Title: A Prospective Multicenter Study on HIV-associated Hodgkin Lymphoma
Brief Title: Prospective Study on HIV-related Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harlachinger Krebshilfe e.V. (Other)
Collaborators: Deutsche AIDS Gesellschaft e.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-HL 2004
Record Dates: First submitted 2011-11-01; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: HIV-associated Hodgkin Lymphoma
MeSH Terms: interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine; Etoposide; Cyclophosphamide; Vincristine; Procarbazine; Prednisone

INTERVENTIONS:
Drug: Doxorubicin — The four-drug ABVD chemotherapy regimen and the seven-drug BEACOPP-baseline chemotherapy regimen contain doxorubicin.
  * Early stage favorable Hodgkin Lymphoma: 2 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) + 30 Gy involved field (IF) radiation
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of ABVD + 30 Gy involved field (IF) radiation or 4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP)-baseline + 30 Gy IF radiation
  * Advanced Hodgkin Lymphoma: 8 cycles of BEACOPP-baseline. After the completion of chemotherapy sites of initial bulky disease (those at least 5 cm in diameter) and residual tumor larger than 2.5 cm in diameter receive 30 Gy of irradiation.
Drug: Bleomycin — The four-drug ABVD chemotherapy regimen and the seven-drug BEACOPP-baseline chemotherapy regimen contain bleomycin.
  * Early stage favorable Hodgkin Lymphoma: 2 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) + 30 Gy involved field (IF) radiation
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of ABVD + 30 Gy involved field (IF) radiation or 4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP)-baseline + 30 Gy IF radiation
  * Advanced Hodgkin Lymphoma: 8 cycles of BEACOPP-baseline. After the completion of chemotherapy sites of initial bulky disease (those at least 5 cm in diameter) and residual tumor larger than 2.5 cm in diameter receive 30 Gy of irradiation.
Drug: Vinblastine — The four-drug ABVD chemotherapy regimen contains vinblastine
  * Early stage favorable Hodgkin Lymphoma: 2 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) + 30 Gy involved field (IF) radiation
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of ABVD + 30 Gy involved field (IF) radiation
Drug: Dacarbazine — The four-drug ABVD chemotherapy regimen contains dacarbazine
  * Early stage favorable Hodgkin Lymphoma: 2 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) + 30 Gy involved field (IF) radiation
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of ABVD + 30 Gy involved field (IF) radiation
Drug: Etoposide — The seven-drug BEACOPP-baseline chemotherapy regimen contains etoposide.
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP)-baseline + 30 Gy IF radiation
  * Advanced Hodgkin Lymphoma: 8 cycles of BEACOPP-baseline. After the completion of chemotherapy sites of initial bulky disease (those at least 5 cm in diameter) and residual tumor larger than 2.5 cm in diameter receive 30 Gy of irradiation.
Drug: Cyclophosphamide — The seven-drug BEACOPP-baseline chemotherapy regimen contains cyclophosphamide.
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP)-baseline + 30 Gy IF radiation
  * Advanced Hodgkin Lymphoma: 8 cycles of BEACOPP-baseline. After the completion of chemotherapy sites of initial bulky disease (those at least 5 cm in diameter) and residual tumor larger than 2.5 cm in diameter receive 30 Gy of irradiation.
Drug: Vincristine — The seven-drug BEACOPP-baseline chemotherapy regimen contains vincristine.
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP)-baseline + 30 Gy IF radiation
  * Advanced Hodgkin Lymphoma: 8 cycles of BEACOPP-baseline. After the completion of chemotherapy sites of initial bulky disease (those at least 5 cm in diameter) and residual tumor larger than 2.5 cm in diameter receive 30 Gy of irradiation.
Drug: Procarbazine — The seven-drug BEACOPP-baseline chemotherapy regimen contains procarbazine.
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP)-baseline + 30 Gy IF radiation
  * Advanced Hodgkin Lymphoma: 8 cycles of BEACOPP-baseline. After the completion of chemotherapy sites of initial bulky disease (those at least 5 cm in diameter) and residual tumor larger than 2.5 cm in diameter receive 30 Gy of irradiation.
Drug: Prednisone — The seven-drug BEACOPP-baseline chemotherapy regimen contains prednisone.
  * Early stage unfavorable Hodgkin Lymphoma: 4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP)-baseline + 30 Gy IF radiation
  * Advanced Hodgkin Lymphoma: 8 cycles of BEACOPP-baseline. After the completion of chemotherapy sites of initial bulky disease (those at least 5 cm in diameter) and residual tumor larger than 2.5 cm in diameter receive 30 Gy of irradiation.

SUMMARY:
Standard therapy for HIV-related Hodgkin lymphoma (HIV-HL) has not been defined. This trial was initiated to investigate a risk adapted treatment strategy in patients (pts) with HIV-HL as established in HIV-negative patients with HL.

Treatment schedule:

* Early stage favorable Hodgkin Lymphoma (HL): 2 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) plus 30 Gy involved field (IF) radiation
* Early stage unfavorable HL: 4 cycles of bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPP)-baseline or 4 cycles of ABVD plus 30 Gy IF radiation
* Advanced HL: 8 cycles of BEACOPP-baseline. BEACOPP should be replaced by ABVD in pts with far advanced HIV-infection. After the completion of chemotherapy sites of initial bulky disease (those at least 5 cm in diameter) and residual tumor larger than 2.5 cm in diameter receive 30 Gy of irradiation.
* Primary outcome measure: tolerability, treatment-related mortality
* Secondary outcome measure: complete remission rate, progression-free survival (PFS), overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 75 years
* proven infection with HIV 1 (Elisa and Western Blot)
* histology-proven newly diagnosed Hodgkin lymphoma
* written, informed consent.

Exclusion Criteria:

* severe cardiac, hepatic or pulmonary insufficiency
* severe renal insufficiency (creatinine > 2,0 mg/dl) not caused by lymphoma
* bone marrow failure, not caused by lymphoma or HAART (neutrophils < 1000/µl, platelets < 70.000/µl)
* uncontrolled infection
* uncontrolled drug addiction or psychiatric disease
* pregnancy or lactation period
* prior chemotherapy of Hodgkin lymphoma
* life expectancy < 6 weeks
* HIV-related wasting-syndrome
* active secondary malignancy with cervix carcinoma in situ, basalioma and Kaposi's sarcoma being excepted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2004-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with World Health Organization (WHO) grade 3 and grade 4 toxicity | 30 days after termination of chemotherapy or radiotherapy
Treatment related mortality | 30 days after termination of chemotherapy or radiotherapy

SECONDARY OUTCOMES:
Overall Survival | 12 months and 24 months after termination of chemotherapy or radiotherapy
Progression-free survival | 12 months and 24 months after termination of chemotherapy or radiotherapy
Complete remission rate | 30 days and 90 days after termination of chemotherapy or radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hentrich, MD, Principal Investigator — Harlaching Hospital, Academic Teaching Hospital of the University of Munich, Department of Hematology, Oncology and Palliative Care
Locations (8):
- Germany (8):
  - Vivantes Auguste Victoria Klinikum, Berlin
  - Ärzteforum Seestrasse, Berlin
  - Universiy of Bonn, Bonn
  - University of Cologne, Cologne
  - University of Frankfurt, Frankfurt
  - Asklepios Klinikum St. Georg, Hamburg
  - Infektionsmedizinisches Zentrum Hamburg, Hamburg
  - Harlaching Hospital, Munich